CLINICAL TRIAL: NCT00274976
Title: Subcutaneous Campath-1H in Fludarabine-Refractory CLL
Brief Title: Alemtuzumab in Treating Patients With Advanced Chronic Lymphocytic Leukemia That Did Not Respond to Previous Fludarabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455059; GCLLSG-CLL2H; EU-20550; MEDAC-GCLLSG-CLL2H; AMGEN-GCLLSG-CLL2H
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2006-05

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

INTERVENTIONS:
Biological: alemtuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This phase II trial is studying how well giving alemtuzumab by injection works in treating patients with advanced chronic lymphocytic leukemia that did not respond to previous fludarabine.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and efficacy of subcutaneous alemtuzumab vs intravenous alemtuzumab in patients with fludarabine-refractory advanced chronic lymphocytic leukemia.
* Determine the response in patients with high-risk genetic abnormalities (unmutated immunoglobulin variable heavy-chain [IgVH] status, del [17p], del [11q]) treated with subcutaneous alemtuzumab after progression on fludarabine.

OUTLINE: This is a multicenter study.

Patients receive alemtuzumab IV once, followed 1 week later by alemtuzumab subcutaneously once weekly for up to 12 weeks.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of previously treated advanced chronic lymphocytic leukemia (CLL)

  * Fludarabine-refractory disease
  * Requires treatment

PATIENT CHARACTERISTICS:

* Life expectancy more than 6 months
* ECOG 0-2
* No severe organ dysfunction
* No other concomitant or previous neoplasms
* No autoimmune hemolytic anemia or thrombocytopenia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Up to 5 prior chemotherapy regimens allowed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy
Response

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Stilgenbauer, MD — Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm
Locations (35):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Germany (34):
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - Specialist Practice for Oncology, Aschaffenburg
  - Humaine - Clinic, Bad Saarow
  - Haematolo-Onkologische Schwerpunktpraxis - Berlin, Berlin
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Hospital Kuchwald Chemnitz, Chemnitz
  - Universitaetsklinikum Essen, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - Praxis fur Innere Medizin - Hamburg, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Marienhospital at Ruhr University Bochum, Herne
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Internistische Praxis - Landshut, Landshut
  - Klinikum Lippe - Lemgo, Lemgo
  - III Medizinische Klinik Mannheim, Mannheim
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Klinikum Oldenburg, Oldenburg
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - Medizinische Klinik und Poliklinik II - Universitaetsklinikum Wuerzburg, Würzburg

REFERENCES:
- [Result] Stilgenbauer S, Zenz T, Winkler D, Buhler A, Schlenk RF, Groner S, Busch R, Hensel M, Duhrsen U, Finke J, Dreger P, Jager U, Lengfelder E, Hohloch K, Soling U, Schlag R, Kneba M, Hallek M, Dohner H; German Chronic Lymphocytic Leukemia Study Group. Subcutaneous alemtuzumab in fludarabine-refractory chronic lymphocytic leukemia: clinical results and prognostic marker analyses from the CLL2H study of the German Chronic Lymphocytic Leukemia Study Group. J Clin Oncol. 2009 Aug 20;27(24):3994-4001. doi: 10.1200/JCO.2008.21.1128. Epub 2009 Jul 13. PMID 19597025
- [Result] Zenz T, Habe S, Denzel T, Mohr J, Winkler D, Buhler A, Sarno A, Groner S, Mertens D, Busch R, Hallek M, Dohner H, Stilgenbauer S. Detailed analysis of p53 pathway defects in fludarabine-refractory chronic lymphocytic leukemia (CLL): dissecting the contribution of 17p deletion, TP53 mutation, p53-p21 dysfunction, and miR34a in a prospective clinical trial. Blood. 2009 Sep 24;114(13):2589-97. doi: 10.1182/blood-2009-05-224071. Epub 2009 Jul 30. PMID 19643983
- [Result] Stilgenbauer S, Zenz T, Winkler D, et al.: Subcutaneous alemtuzumab (Campath) in fludarabine-refractory CLL: final results of the CLL2H trial of the GCLLSG and comprehensive analysis of prognostic markers. [Abstract] Blood 112 (11): A-329, 2008.
- [Derived] Schnaiter A, Paschka P, Rossi M, Zenz T, Buhler A, Winkler D, Cazzola M, Dohner K, Edelmann J, Mertens D, Kless S, Mack S, Busch R, Hallek M, Dohner H, Stilgenbauer S. NOTCH1, SF3B1, and TP53 mutations in fludarabine-refractory CLL patients treated with alemtuzumab: results from the CLL2H trial of the GCLLSG. Blood. 2013 Aug 15;122(7):1266-70. doi: 10.1182/blood-2013-03-488197. Epub 2013 Jul 2. PMID 23821658